CLINICAL TRIAL: NCT06575218
Title: The Effectiveness of Virtual Reality Training Program in Community Dwelling Older Adults With Alzheimer's Disease
Brief Title: The Effectiveness of Virtual Reality Training Program
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yeditepe University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: YeditepeUni
Record Dates: First submitted 2024-08-23; First posted 2024-08-28 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Virtual reality training group (Experimental): It will be included in the virtual reality training program to be implemented with the Wii-fit console.
  Interventions: Other: Conventional exercise and cognitive exercise; Other: control
- Conventional exercise and cognitive exercise group (Experimental): It will be included in the cognitive exercise program along with conventional balance exercises.
  Interventions: Device: Virtual reality training; Other: control
- Control group (No Intervention): no intervention

INTERVENTIONS:
Device: Virtual reality training — Virtual reality training
  Arms: Conventional exercise and cognitive exercise group
Other: Conventional exercise and cognitive exercise — Conventional exercise and cognitive exercise
  Arms: Virtual reality training group
Other: control — no intervention
  Arms: Conventional exercise and cognitive exercise group; Virtual reality training group

SUMMARY:
Alzheimer's disease is the most common type of dementia, accounting for 50% of all cases. Advanced age is a significant risk factor for AD. Virtual Reality (VR) is an interactive video game technology that provides computer-generated environments that include physical activity and provide users with experiences similar to those in the real world. VR technology can be used for rehabilitation purposes in individuals with various orthopedic and neurological disorders due to its ability to enhance motor, cognitive learning and neural plasticity (1,2). The aim of our study was to examine the effect of the Virtual Reality Training Program on cognition in individuals with Alzheimer's disease living in the community.

DETAILED DESCRIPTION:
The aim of our study was to examine the effect of the Virtual Reality Training Program on cognition in individuals with Alzheimer's disease living in the community. Prospective Randomized Controlled Single Blind Study After the patients and their relatives are informed in detail before the study, they will be asked whether they want to participate in the study and the individuals or relatives of the patients who approve of participating in the study will be asked to sign the informed consent form. Individuals who meet the inclusion criteria will be randomly divided into three groups by a single researcher: Virtual reality training program, cognitive exercise with traditional balance exercises, and traditional balance exercises only.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 55 years and older Diagnosed with AD according to DSM-IV diagnostic criteria by a neurologist, MOCA ≥ 16 Clinical Dementia Rating Scale < 2

Exclusion Criteria:

* Various mobility restrictions, musculoskeletal disorders, (wheelchair use, etc.) Clinically significant aphasia (must be able to understand the therapist's commands) Significant visual or sensory impairment

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-05-21 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-09-06 (Estimated)

PRIMARY OUTCOMES:
Montreal cognitive assessment scale | 12 weeks
  MOCA is a short cognitive assessment method developed to detect particularly mild stages of cognitive impairment.
Berg Balance Scale | 12 weeks
  BBS measures static and dynamic balance in elderly individuals
Time up and Go Test | 12 weeks
  TUG test evaluates fall risk, mobility and physical performance in the elderly

CONTACTS AND LOCATIONS:
Locations (1):
- Ebru Akbuğa Koç, Istanbul, Turkey (Türkiye)